CLINICAL TRIAL: NCT04870060
Title: A Pharmacokinetic-pharmacodynamic Study Assessing the Ability of Curcumin to Decrease Cytokines Involved in Mucositis in the Autologous Transplant Setting
Brief Title: Ability of Curcumin to Decrease Cytokines Involved in Mucositis in the Autologous Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Navin Khattry, Professor and BMT convener, Tata Memorial Centre
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 641
Record Dates: First submitted 2021-04-17; First posted 2021-05-03 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2021-04

CONDITIONS: Oral Mucositis (Ulcerative)
Keywords: Curcumin; Cytokines; Mucositis; Autologous HSCT; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Stomatitis; Ulcer; Mucositis

STUDY DESIGN:
Intervention Model Description: prospective, single centre, pilot pharmacokinetic and pharmacodynamic study with an adaptive design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in this arm received only standard supportive care
- Curcumin (Experimental): Patients in this arm received curcumin lozenges (4 lozenges BD) along with standard supportive care
  Interventions: Drug: Curcumin Lozenges

INTERVENTIONS:
Drug: Curcumin Lozenges — Curcumin lozenges - 4 lozenges to be chewed BD. Each lozenge contained 100 mg of curcumin and the formulation was Solid Lipid Curcumin Particle (SLCP)
  Other Names: Longvida (Pharmanza Herbal Pvt Ltd.)
  Arms: Curcumin

SUMMARY:
Mucositis is a very common complication in bone marrow transplant setting. It is a result of injury to the gut caused by high dose chemotherapy. Currently there are no universal protocols that have been accepted as a standard to prevent and treat mucositis in the transplant setting. Post transplant upto 80% of patients suffer from a severe mucositis. Proinflammatory cytokines play a major role in the development of mucositis. Interventions that decrease the levels of these cytokines may be beneficial in preventing mucositis. This study is aimed at evaluating the role of curcumin in reducing cytokine levels and the incidence and duration of mucositis in patients undergoing autologous stem cell transplantation.

DETAILED DESCRIPTION:
Mucositis is an inevitable side-effect of intensive conditioning therapy used for hematopoietic stem cell transplantation and usually refers to the mucosal ulceration of mouth and throat. However, it is generally accepted that oral mucositis (OM) is in reality the most obvious manifestation of damage or injury elsewhere particularly that of the gut. The incidence of oral mucositis (WHO grades I-IV ) with certain myeloablative conditioning regimens has been reported in up to 90% with range of severe mucositis (WHO grade III/IV) from 10 to 78%.

Mucositis is a complex biological process which occurs in four phases - 1. inflammatory/vascular phase; 2. epithelial phase; 3. ulcerative/bacteriological phase; 4. healing phase. Each phase is interdependent and is the consequence of a series of actions mediated by cytokines, the direct effect of the chemotherapeutic drug on the epithelium, the oral bacterial flora and the status of the patient's bone marrow. Pro-inflammatory cytokines such as interleukin -1 (IL-1), interleukin -6 (IL-6),interleukin-8 (IL-8), interleukin-17 (IL-17), Tumour Necrosis Factor-alpha (TNF-α), Transforming Growth Factor-B (TGF-B),Interferon gamma (IFN-γ) and certain prostaglandins play a central role in its pathogenesis. Chemotherapy, in particular, affects the release of both interleukin-1 (IL-1) and tumor necrosis factor-alpha (TNF-α)from the epithelium. TNF-α is capable of causing tissue damage and may be an accelerating and initiating event in the mucositis process. IL-1 incites an inflammatory response resulting in increased sub-epithelial vascularity with a potential consequent increase in the local levels of cytotoxic agent. On the other hand, cytokines like TGF-β are known inhibitors of epithelial cell proliferation by preventing cell cycle progression and accumulating cells in G1 or G0. For clonogenic stem cells in the intestine, this might render them more resistant to the cytotoxic damage, leaving more clonogenic stem cells to start the regeneration process. Cytokine modulation is the primary mechanism of action of several agents experimented in the recent past to reduce mucositis. For example, Triclosan oral rinse and interleukin-11 (IL-11) therapy reduce ulceration and duration of mucositis by downregulation of PGE2, TNF-α, IL-12 and IFN-γ. It is quite possible that a role exists for transcription factors which modify the genetic expression of cytokines and enzymes which are critical in producing tissue damage. Such factors, such as NF-kappa B, increase the rate of gene transcription and thereby the rate of messenger RNA and protein production. Therefore inhibition of NF-kB could be beneficial in the reduction of mucosal injury.

Currently there are no universal protocols that have been accepted as a standard to prevent and treat OM in the transplant setting. Research is proceeding on several new fronts. Palifermin, recombinant human - keratinocyte growth factor-1, has been shown to the most effective agent so far in few phase II studies.

Accumulating evidence suggests that curcumin inhibits various inflammatory cytokines through inhibition of Nuclear Factor Kappa- β. Curcumin, polyphenol derivative with low toxicity profile, is commonly used in India for its anti-inflammatory actions. It is derived from the plant Curcuma longa. In vitro studies have shown potent anti-inflammatory activity at concentrations of 1 umol/L. Though oral bioavailability of curcumin is poor, in vivo sepsis models in mice have shown good anti-inflammatory activity despite poor plasma levels. Similarly significant decrease of ex vivo production of LPS induced PGE2 levels have been seen in patients treated with curcumin.

Phase I studies in cancer patients have shown that curcumin can be given at doses ranging from 440 mg to 12 grams daily without any toxicity. There was no dose-limiting toxicity; dosing was limited by the number of pills that patients could or would swallow daily. Curcumin used for cancer prevention is seldom administered in a pure chemical form. Rather, it typically consists of three separate curcuminoids consisting of curcumin itself as well as demethoxycurcumin and bisdesmethoxycurcumin. Plasma levels of curcumin and its metabolites such as curcumin glucuronide and curcumin sulphate have been shown to be in the range of 10- 50 ng/ml in patients receiving doses greater than 3.6 gms daily. This peak concentration is seen 1 hour after a given dose. In a recently published study of curcumin in pancreatic cancer little, if any, free or unconjugated curcumin was detected in the plasma of 19 subjects who received a daily dose of 8 g curcumin. An apparent steady-state level of conjugated curcumin in plasma that was achieved by day 3; this level was 22 to 41 ng/mL. Though the peak plasma concentration of curcumin detected is low, at these doses, biological activity demonstrated by either reduction of cytokine levels or decrease in the activity of NK-kB has been seen in all patients.

There are no studies exploring the role of curcumin in mucositis in patients undergoing high dose chemotherapy .The Investigators aim to study the pharmacokinetics and pharmacodynamics of curcumin in the above setting. Patients with mucositis may have difficulty in swallowing tablets. Therefore a lozenge formulation of curcumin will be employed in this study. Lozenges will be manufactured by Pharmanza Herbal Pvt. Ltd (PH). Each lozenge of 1g contains 100mg of curcumin. A capsule formulation of curcumin manufactured by PH containing 27% of curcuminoids was employed in an earlier study in osteogenic sarcoma patients at this centre. Single dose pharmacokinetics with 4g of the formulation yielded peak curcumin concentration of 37.69 ng/ml and half-life of about 2.5 hours - (unpublished data). The time to peak concentration was around 3 hours. Based on this data, a dose of four lozenges (4 gm) twice a day (BID) was deemed necessary and sufficient to achieve the desired inhibition of NF-kB.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years and above .
2. Patients who give written informed consent
3. Patients with performance status - 0,1 or 2(ECOG scale)
4. Patients receiving any of the following high dose chemotherapy regimens

   1. Melphalan- 200 mg/m2 or more (MEL-200 mg/m2)
   2. Busulfan and Melphalan (BuMEL)
   3. Carmustine (BCNU), Etoposide, Cytosine Arabinoside and Melphalan ( BEAM)
5. Patients who have creatinine clearance > 50 ml/min
6. Patients with serum bilirubin levels < 2mg/dl. and serum liver enzymes (ALT or AST or both) greater than 5 times the upper limit of normal value.

Exclusion Criteria:

1. Patients who are on NSAIDs , aspirin ,antioxidants or systemic steroids for more than 3 months and the last dose taken within the last one week.
2. Patients being treated for active infection at the time of starting high dose chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10-06 (Actual); Primary Completion 2015-07-03 (Actual); Study Completion 2015-07-03 (Actual)

PRIMARY OUTCOMES:
Serum TNF alpha AUC (0-28) | Day+28
  This will be calculated using serum TNF alpha levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Salivary TNF alpha AUC (0-28) | Day+28
  This will be calculated using salivary TNF alpha levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Serum Interleukin 1 AUC (0-28) | Day+28
  This will be calculated using serum IL-1 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Salivary Interleukin 1 AUC (0-28) | Day+28
  This will be calculated using salivary IL-1 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Serum Interleukin 6 AUC (0-28) | Day+28
  This will be calculated using serum IL-6 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Salivary Interleukin 6 AUC (0-28) | Day+28
  This will be calculated using salivary IL-6 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Serum Interleukin 8 AUC (0-28) | Day+28
  This will be calculated using serum IL-8 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Salivary Interleukin 8 AUC (0-28) | Day+28
  This will be calculated using salivary IL-8 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Serum Interleukin 17 AUC (0-28) | Day+28
  This will be calculated using serum IL-17 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Salivary Interleukin 17 AUC (0-28) | Day+28
  This will be calculated using salivary IL-17 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Serum TGF-beta AUC (0-28) | Day+28
  This will be calculated using serum TGF-beta levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Salivary TGF-beta AUC (0-28) | Day+28
  This will be calculated using salivary TGF-beta levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Serum Interferon gamma AUC (0-28) | Day+28
  This will be calculated using serum IFN-gamma levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Salivary Interferon gamma AUC (0-28) | Day+28
  This will be calculated using salivary IFN-gamma levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Serum Prostaglandin E2 AUC (0-28) | Day+28
  This will be calculated using serum prostaglandin E2 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Salivary Prostaglandin E2 AUC (0-28) | Day+28
  This will be calculated using salivary prostaglandin E2 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14 and then on day+28. Using these values, AUC (0-28) will be calculated using linear trapezoidal model
Plasma curcumin AUC (0-12 hr) | Up to 12 hours from 1st dose
  This will be done using plasma curcumin levels measured 1 hour prior to the first dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 (± 15 min) hours post dose.
Plasma Bis-demethoxycurcumin AUC (0-12 hr) | Up to 12 hours from 1st dose
  This will be done using plasma Bis-demethoxycurcumin levels measured 1 hour prior to the first dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 (± 15 min) hours post dose.
Plasma demethoxycurcumin AUC (0-12 hr) | Up to 12 hours from 1st dose
  This will be done using plasma demethoxycurcumin levels measured 1 hour prior to the first dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 (± 15 min) hours post dose.

SECONDARY OUTCOMES:
Mucositis incidence | Till hospital discharge or till day+28 (whichever is earlier)
  To evaluate the incidence of grade 3 or 4 (WHO) oral mucositis on patients taking oral curcumin in post autologous transplant setting.
Mucositis duration | Till hospital discharge or till day+28 (whichever is earlier)
  To evaluate the duration of grade 3 or 4 (WHO) oral mucositis on patients taking oral curcumin in post autologous transplant setting.
Diarrhoea incidence | Till hospital discharge or till day+28 (whichever is earlier)
  To evaluate the incidence of grade 3 or 4 (CTCAE v 3.0) diarrhea on patients taking oral curcumin in post autologous transplant setting.
Diarrhoea duration | Till hospital discharge or till day+28 (whichever is earlier)
  To evaluate the duration of grade 3 or 4 (CTCAE v 3.0) diarrhea on patients taking oral curcumin in post autologous transplant setting.

CONTACTS AND LOCATIONS:
Overall Officials: Navin Khattry, MD, DM, Principal Investigator — Tata Memorial Centre
Locations (1):
- Tata Memorial Centre, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Punatar S, Katti K, Rajamanickam D, Patil P, Dhakan C, Bagal B, Gokarn A, Bonda A, Nayak L, Gurjar M, Kannan S, Chiplunkar S, Gota V, Khattry N. Role of Curcumin in Reducing Toxicities Associated With Mucosal Injury Following Melphalan-Based Conditioning in Autologous Transplant Setting. Cell Transplant. 2022 Jan-Dec;31:9636897221086969. doi: 10.1177/09636897221086969. PMID 35435039